CLINICAL TRIAL: NCT03765554
Title: A PHASE 1, OPEN-LABEL STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE PHARMACOKINETICS OF PF-06700841 FOLLOWING SINGLE ORAL ADMINISTRATION OF MODIFIED RELEASE TABLETS COMPARED TO IMMEDIATE RELEASE TABLETS UNDER FASTED CONDITIONS
Brief Title: Clinical Study to Evaluate Blood Concentrations of PF-06700841 After Oral Dose as Different Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7931010; 2018-003512-41 (EudraCT Number)
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — PF-06700841

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PF-06700841: IR followed by MR (Experimental): Participants receive PF-06700841 Immediate release tablets (IR) followed by PF-06700841 Modified release tablets (MR)
  Interventions: Drug: PF-06700841 Immediate release tablets; Drug: PF-06700841 Modified release tablets
- PF-06700841: MR followed by IR (Experimental): Participants receive PF-06700841 Modified release tablets (MR) followed by PF-06700841 Immediate release tablets (IR)
  Interventions: Drug: PF-06700841 Immediate release tablets; Drug: PF-06700841 Modified release tablets

INTERVENTIONS:
Drug: PF-06700841 Immediate release tablets — Small molecule tablets in immediate release form
Drug: PF-06700841 Modified release tablets — Small molecule tablets in modified release form

SUMMARY:
PF-06700841 is a dual Tyrosine kinase 2 (TYK2) Janus kinase 1 (JAK1) inhibitor that is being developed for oral treatment of adult patients with Inflammatory Bowel Disease (IBD).This open-label study will evaluate the pharmacokinetics of PF-06700841 following single oral doses of immediate release (IR) and modified release (MR) tablets in healthy, adult participants under fasted conditions. This is an open label, single dose, randomized, 2 period, 2- sequence crossover study in a single cohort of approximately 8 (minimum 6) healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male, and female participants between the ages of 18 and 55 years at the time of screening, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Key Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Have or have had clinically significant infections within the past 3 months prior to the first dose of investigational product (eg, those requiring hospitalization or parenteral antibiotics, or as judged by the Investigator), evidence of any infection within the past 7 days prior to the first dose of investigational product, herpes simplex within 12 weeks or history of disseminated herpes simplex infection, symptomatic herpes zoster or recurrent (>1 episode) or disseminated herpes zoster.
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb) or hepatitis C antibody (HCVAb). As an exception, a positive hepatitis B surface antibody (HepBsAb) finding as a result of participant vaccination is permissible.
* History of tuberculosis or active or latent or inadequately treated infection, positive QuantiFERON tuberculosis (TB) Gold test.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product used in this study (whichever is longer).
* Female participants who are pregnant or wish to become pregnant; breastfeeding females.
* Males/Females of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-06700841 | pre-dose, 1,2,4,6,8,10,12,16,24,28,32,36,48 hour post-dose
Area under the plasma concentration-time curve from time zero to the last measured concentration (AUClast) of PF-06700841 | pre-dose, 1,2,4,6,8,10,12,16,24,28,32,36,48 hour post-dose
Time to reach maximum observed plasma concentration (Tmax) of PF-06700841 | pre-dose, 1,2,4,6,8,10,12,16,24,28,32,36,48 hour post-dose
Area under the plasma concentration-time curve from time zero to extrapolated infinite time (AUCinf) of PF-06700841 if data permit | pre-dose, 1,2,4,6,8,10,12,16,24,28,32,36,48 hour post-dose

SECONDARY OUTCOMES:
Change from baseline in 12-Lead Electrocardiogram (ECG) parameters - PR interval, QRS complex, QT interval and QTC interval | Pre-dose and 48 hours post-dose
Change from baseline in heart rate | Pre-dose and 48 hours post-dose
Change from baseline in blood pressure | Pre-dose and 48 hours post-dose
Change from baseline in pulse rate | Pre-dose and 48 hours post-dose
Change from baseline in oral temperature | Pre-dose and 48 hours post-dose
Number of participants with laboratory abnormalities | Baseline and 48 hours post-dose
Number of participants with Treatment -Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Discontinuation Due to AEs | Baseline to 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931010&StudyName=A+Phase+1%2C+Open+Label+Study+In+Healthy+Participants+To+Investigate+The+Pharmacokinetics+Of+Pf+06700841+Following+Single+Oral+Administration+Of+Modified+Release+Tablets+Compared+To+Immediate+Release+Tablets+Under+Fasted+Conditions
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7931010&StudyName=A+Phase+1%2C+Open-label+Study+In+Healthy+Participants+To+Investigate+The+Pharmacokinetics+Of+Pf-06700841+Following+Single+Oral+Administration+Of+Modified+Release+Tablets+Compared+To+Immediate+Release+Tablets+Under+Fasted+Conditions